CLINICAL TRIAL: NCT07175649
Title: Methylprednisolone Sodium Succinate With Endovascular ThRombectomy for Large Ischemic STroke: A Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Methylprednisolone Sodium Succinate With Endovascular ThRombectomy for Large Ischemic STroke
Acronym: PEARL-MERIT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYSKY-2025-603-03
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Ischemic Stroke, Acute
MeSH Terms: conditions — Ischemic Stroke | interventions — Methylprednisolone Hemisuccinate; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methylprednisolone group (Experimental)
  Interventions: Drug: Methylprednisolone sodium succinate
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylprednisolone sodium succinate — Intravenous methylprednisolone sodium succinate will be administered at a dose of 2 mg/kg/day for 3 days, with a maximum daily dose of 160 mg (4 vials, 40 mg/vial).
  It is recommended that the initial dose be administered as soon as possible after randomization.
  Other Names: Methylprednisolone
  Arms: Methylprednisolone group
Drug: Placebo — Matched intravenous placebo will be administered for 3 days, with a maximum daily dose of 4 vials.
  Arms: Placebo group

SUMMARY:
It is uncertain whether intravenous methylprednisolone improves outcomes for acute anterior circulation large vessel occlusion (LVO) patients with a large infarct core. In this study, the investigators hypothesize that methylprednisolone plus endovascular thrombectomy (EVT) might be superior to EVT alone in patients with evidence of a large infarct volume. The primary objective of the study is to establish the efficacy of methylprednisolone with EVT in patients with acute anterior circulation LVO and a large infarct core.

DETAILED DESCRIPTION:
The PEARL-MERIT is a multicenter, prospective, randomized, double-blind, placebo-controlled trial. A total of 912 patients (aged 18-85 years) within 24 hours of symptom onset of acute ischemic stroke, who have imaging evidence of an occlusion of the intracranial internal carotid artery (ICA) and/or M1/M2 segment of middle cerebral artery (MCA), a large infarct core, and a planned EVT, will be enrolled.

Patients fulfilling all of the inclusion criteria and none of the exclusion criteria will be randomized 1:1 into 2 groups after obtaining informed consent. One group will receive methylprednisolone, the other group will receive placebo. The primary objective is to evaluate the efficacy of methylprednisolone with EVT compared to placebo with EVT in patients with acute ischemic stroke due to anterior circulation LVO and a large infarct core.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 85 years;
* Clinically diagnosed acute ischemic stroke with screening NIHSS ≥6;
* Time from last known well to randomization ≤24 hours;
* Pre-stroke mRS score of 0-1;
* Occlusion of the responsible vessel confirmed by CT angiography (CTA), magnetic resonance angiography (MRA), or digital subtraction angiography (DSA) in intracranial segment of internal carotid artery (ICA), M1 or M2 segment of middle cerebral artery (MCA), and plan to undergo EVT;
* Alberta Stroke Program Early CT Score (ASPECTS) of 0-5 on NCCT, or ischemic core volume ≥70 mL (defined as regional cerebral blood flow [rCBF] <30% on CT perfusion [CTP] or apparent diffusion coefficient [ADC] <620×10-⁶ mm²/s on MRI);
* Informed consent obtained.

Exclusion Criteria:

* Intracranial hemorrhage on NCCT or MRI;
* Allergy to corticosteroids;
* Allergy to contrast agents;
* Severe infectious disease unsuitable for corticosteroid therapy or concurrent contraindications to corticosteroid treatment;
* Random blood glucose >22.2 mmol/L (400 mg/dL);
* Known hereditary or acquired bleeding diathesis, coagulation factor deficiency, use of warfarin with an international normalized ratio (INR) >1.7, or administration of novel oral anticoagulants within 48 hours of symptom onset;
* Platelet count <90×10⁹/L;
* History of gastrointestinal or urinary tract bleeding within the last month;
* Current participation in another interventional clinical trial;
* Pregnancy or lactating;
* Renal dysfunction with an estimated glomerular filtration rate (eGFR) <30 mL/min or serum creatinine >220 μmol/L (2.5 mg/dL);
* Persistent systolic blood pressure >185 mmHg or diastolic blood pressure >110 mmHg despite antihypertensive treatment;
* Life expectancy <6 months due to terminal illnesses such as malignancy or severe cardiopulmonary disease;
* Intracranial aneurysm or arteriovenous malformation;
* Intracranial tumour with mass effect on imaging (except for small meningiomas);
* Other conditions deemed unsuitable for study participation by the investigator, including inability to comprehend and/or comply with study procedures and/or follow-up due to psychiatric, cognitive, or emotional disorders.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 912 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
The modified Rankin Scale score (mRS) 0-3 | 90±14 days after randomization
  The proportion of mRS score 0-3 at 90 (±14) days

SECONDARY OUTCOMES:
The distribution of the modified Rankin Scale scores | 90±14 days after randomization
  The shift analysis of mRS at 90±14 days (merged 0-1)
The modified Rankin Scale score (mRS) 0-4 | 90±14 days after randomization
  The proportion of mRS score 0-4 at 90 (±14) days
The modified Rankin Scale score (mRS) 0-2 | 90±14 days after randomization
  The proportion of mRS score 0-2 at 90 (±14) days
The modified Rankin Scale score (mRS) 0-1 | 90±14 days after randomization
  The proportion of mRS score 0-1 at 90 (±14) days
Quality of Life (EQ-5D-5L) | 90±14 days after randomization
  Quality of life measured by EQ-5D-5L scale score at 90 (±14) days
Neurologic deficit (NIHSS score) changes | 7±1 days after randomization/at discharge
  National Institutes of Health Stroke Scale (NIHSS) score change from baseline, at 7 (±1) days or at discharge
Infarct core volume changes | 7±1 days after randomization/at discharge or at 36±12 hours after randomization
  Infarct core volume change from baseline, assessed with NCCT at 7±1 days after randomization/at discharge or with MRI at 36±12 hours
Rate of decompressive craniectomy | 7±1 days after randomization
  Rate of decompressive craniectomy at 7 (±1) days

OTHER OUTCOMES:
SAFETY OUTCOME: Mortality | 90±14 days after randomization
  All-cause mortality within 90 days
SAFETY OUTCOME: Symptomatic intracranial hemorrhage (sICH) | Within 48 hours after randomization
  Symptomatic intracranial hemorrhage (sICH) within 48 hours (according to Heidelberg criteria)
SAFETY OUTCOME: Any serious adverse events and steroid-related adverse events (hyperglycemia, infection, and gastrointestinal hemorrhage) | 90±14 days after randomization
  Safety will be assessed according to common terminology criteria for adverse events (CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: Yamei Tang, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No